CLINICAL TRIAL: NCT03131531
Title: Bergamo Lymphoid Cancer Registry
Status: Recruiting | Type: Observational
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Principal Investigator, Rambaldi Alessandro, Prof., A.O. Ospedale Papa Giovanni XXIII
Other Study IDs: BLCR
Record Dates: First submitted 2017-04-20; First posted 2017-04-27 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Hodgkin Lymphoma; Non Hodgkin Lymphoma; Myeloma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Biological specimens include peripheral blood, serum, plasma, bone marrow, lymph node, normal or disease-infiltrated tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hodgkin lymphoma
  Interventions: Other: Patient registry
- Non-Hodgkin lymphoma
  Interventions: Other: Patient registry
- Myeloma
  Interventions: Other: Patient registry

INTERVENTIONS:
Other: Patient registry — Clinical data, specific procedures and treatments will follow the Institutional standard operative procedures

SUMMARY:
This registry has been established to gain a better understanding of the clinical and biological characteristics and outcome of patients with lymphoid cancer

DETAILED DESCRIPTION:
Lymphoid cancer including Hodgkin disease, non-Hodgkin lymphomas (NHL) and myeloma, represents the most common hematologic malignancy. Despite the overall prognosis improved in the last 10 years, there are many open issues that need to be addressed, specifically refractoriness to standard treatment, disease recurrence and outcome with new drug in the so called "real world" setting. Since the Hematology and Bone Marrow Transplant Unit at "Ospedale Papa Giovanni XIII" of Bergamo has developed specific tools to collect clinical data thought fully validated electronic charts and biological specimens thanks to a regulatory compliant biobanking program, the aim of this study is to collect clinical and biological information of lymphoid cancer patients. The cohort of patients enrolled will permit to analyze the practice pattern, perform biological correlative studies of great translational potential with relevance to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older
* Written informed consent
* Confirmed diagnosis of Hodgkin disease, non-Hodgkin lymphomas or myeloma

Exclusion Criteria:

- Unconfirmed diagnosis of Hodgkin disease, non-Hodgkin lymphomas or myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for this study are patients with a diagnosis of lymphoid cancer in charge of the Hematology and Bone Marrow Transplant Unit "Ospedale Papa Giovanni XIII" of Bergamo.
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2017-03-23 (Actual); Primary Completion 2027-03-23 (Estimated); Study Completion 2037-03-23 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 20 years
  Analyzed for all patients as time from diagnosis to death as a result of any cause, stratified according to intervention and baseline characteristics

SECONDARY OUTCOMES:
Disease-free survival | 20 years
  Analyzed only for patients in complete response, as time from achievement of the complete response to relapse or death due to disease or acute toxicity of treatment, stratified according to intervention and baseline characteristics
Progression-free survival | 20 years
  Analyzed for all patients, as time from diagnosis to progression of disease or death as a result of any cause, stratified according to intervention and baseline characteristics
Biological correlative studies | 20 years
  Association between clinical and biologic characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Rambaldi, MD, Principal Investigator — A.O. Ospedale Papa Giovanni XXIII
Locations (1):
- Hematology and Bone Marrow Transplant Unit, A.O. Ospedale Papa Giovanni XXIII, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No